CLINICAL TRIAL: NCT03968224
Title: Effectiveness of the Treatment With Dapagliflozin and Metformin Compared to Metformin Monotherapy for Weight Loss on Diabetic and Prediabetic Patients With Obesity Class III
Brief Title: Effectiveness of Dapagliflozin for Weight Loss
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centro Medico Nacional Siglo XXI IMSS (Other)
Responsible Party: Principal Investigator, Aldo Ferreira Hermosillo, Research Associate, Centro Medico Nacional Siglo XXI IMSS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2016-785-094
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: PreDiabetes; Obesity, Morbid; Diabetes Mellitus, Type 2
Keywords: Metformin; Sodium-Glucose Transporter 2 Inhibitors; PreDiabetes; Obesity, Morbid; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Prediabetic State; Obesity, Morbid; Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin/Dapagliflozin (Experimental): Metformin 1,700 mg/day and Dapagliflozin 10 mg/day for a year.
  Interventions: Drug: Dapagliflozin/Metformin
- Metformin (Active Comparator): Metformin 1,700 mg/day
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Dapagliflozin/Metformin — Two tablets of Metformin 850 mg every 12 hours were provided in combination with Dapagliflozin 10 mg per day. Each participant received diet and exercise intervention according to their BMI and current physical condition.
  Other Names: Group 1
  Arms: Metformin/Dapagliflozin
Drug: Metformin — Two tablets of Metformin 850 mg every 12 hours were provided. Each participant received diet and exercise intervention according to their BMI and current physical condition.
  Other Names: Group 2
  Arms: Metformin

SUMMARY:
Mexico has one of the highest prevalence of obesity, reported on 32.4 percent of people over 20 years old, with a prevalence of obesity class III of 1.8 percent on males and 4.1 percent on females.

According to previous data in our Obesity Clinic the mean age of these patients is 41 years, 46 percent have pre-diabetes or type 2 diabetes mellitus (T2D); 66 percent has hypertension and 33 percent has dyslipidemia. The management of alterations in the glucose metabolism in this unit is made by dietary treatment and with the use of metformin at doses of 1,700 mg/day and/or basal insulin.

Dapagliflozin is a selective SGLT2 inhibitor than has shown a sustained effect on the reduction of glycated hemoglobin at 0.4 to 0.8 percent (initial 7.8 to 8.0 percent). Additionally, due to the induction of glycosuria up to 20 to 85 g/day, it has been calculated that its use induces a caloric deficit at 80 to 340 kcal/day. This has been tested in patients with T2D in which induces a weight loss of 2 to 3 kg and in combination with metformin even a weight loss up to 5.07 kg (-6.21 to 3.93 kg) without regain (at least for 2 years). Furthermore, dapagliflozin decrease systolic blood pressure, increases HDL cholesterol concentrations and decreases triglyceride concentration. The drug product action is independent of the insulin production at pancreas, consequently, it exists a possibility of using the drug product on patients with prediabetes or even on other types of diabetes. Regarding the adverse effects related to its use, it has been described an increase in the risk of genitourinary infections with a low risk for inducing hypoglycemia.

A previous study that included 182 patients with T2D inadequately controlled with metformin assessed the effect of dapagliflozin 10 mg in total weight loss after 24 weeks compared to placebo. It was found a decrease in weight of 2.08 kg (2.8 to 1.31 kg), decrease in waist circumference of 1.52 cm (2.74 to 0.31), decrease in total fat mass assessed with densitometry of 1.48 kg (2.22 to 0.74), decrease of visceral fat mass of 258.4 cm^3 (448.1 to 68.6) and subcutaneous fat of 184.9 cm^3 (359.7 to 10.1). Most of these studies on weight and metabolic control have been performed in patients with obesity class II or I. The aim of this study is to assess if dapagliflozin in combination with metformin is at least 10 percent more effective for weight reduction in comparison with metformin in patients with prediabetes or T2D and obesity grade III.

DETAILED DESCRIPTION:
Methods:

A convenience sampling will be done for patients diagnosed with diabetes or prediabetes according to the American Diabetes Association (ADA) criteria, who assist to the Obesity Clinic and meet the selection criteria. Data from patients that during the study protocol are called to undergo bariatric surgery procedure will be used until the time of surgery (intention-to-treat analysis). The prevalence of comorbidities at baseline and the type and dose of drugs used for treatment will be recorded. Patients will be randomized by a random numbers system generated with a computational software and will be assigned to a group: metformin (1,700 mg/day) or metformin (1,700 mg/day) and dapagliflozin 10 mg. All patients will receive dietary treatment and follow-up during the study by the Nutrition Service. Once assigned to the corresponding group, patients will receive an identification code that will be retained throughout the study. One of the researchers not directly involved in patient care, will assign tablets needed for daily intake for a month and then the number of tablets required for 3 months in a sealed envelope. A run-in period will be used to assess tolerance to treatments. This period will be for a month. At this time patients may notice an increase of uresis and will be instructed to increase fluid intake. Anthropometric and biochemical variables will be recorded baseline and at 1, 3, 6 and 12 months. The determination of glucagon, ghrelin, adiponectin, resistin, interleukin 6 (IL-6) and interleukin 10 (IL-10) will be held on initial appointment and before surgery (depending on the response of each patient). For the determination of these cytokines and peptides, an ELISA kit (Enzyme Linked Immunosorbent Assay) will be used. Adherence to treatment will be evaluated and will consist in consumption of 90 percent of pills granted. The patient will be required to return the drug blister. The registration of adverse events will take place from the start of treatment and throughout the study. Each event will be evaluated by researchers and classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 list. CTCAE considers that an adverse event grade 4 or 5 indicates discontinuation of treatment; grade 3 must be submitted to review by the medical team, and grades 1 or 2 require registration and intervention but not discontinuation of treatment. Adverse events will be recorded in the report sheet. An intention-to-treat analysis will be used if patients require treatment with insulin or sulfonylureas (grade 3 adverse event). They will provide information until the time of its inception. Patients who do not achieve weight loss at one year follow-up, will be discarded to their primary care hospital for continue with dietary recommendations.

Sample Size:

A convenience sample will be performed of patients with obesity class III and prediabetes or diabetes according ADA criteria at Obesity Clinic who meet selection criteria. The sample size was calculated using a mean difference formula with data from Zhang et al. who evaluated weight loss in patients using metformin/dapagliflozin and compared with placebo. Sample size required is 90 patients: 45 patients in metformin group and 45 patients in dapagliflozin/metformin group. Considering a loss of 20 percent of population during study, the final sample size required is 108 patients: 54 patients in metformin and 54 patients in dapagliflozin group.

Statistical analysis Quantitative variables were described using measures of central tendency and dispersion according to the data distributions. Qualitative variables were described using frequencies or percentages. The Shapiro-Wilk test was used to establish normality in the distribution of quantitative variables. Because information on the different quantitative variables was available up to different time periods, a mixed model analysis was performed using the restricted maximum likelihood (REML) method, as well as a mixed model considering the fixed effects of assigned treatment, sex, and prediabetes or diabetes status, and the random effects of variability in weight loss over time. Comparisons between groups were analyzed using Sidak's post-hoc test. Pearson's chi-square test or Fisher's exact test were used to evaluate the association between qualitative variables. Statistical significance was defined as a p < 0.05. Data analysis was performed using SPSS version 17.0 and STATA version 11.0.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than or equal to 40 kg/m^2
* Diagnosis of diabetes or prediabetes according to the criteria of the ADA
* Patients who sign informed consent letter

Exclusion Criteria:

* Use of insulin or sulfonylureas
* Chronic renal failure with glomerular filtration rate <60 ml/min/1.73 m^2
* Use of loop diuretics with no possibility to suspend
* Active genitourinary tract infections determined by symptomatology or urinalysis
* Use of drugs for weight control
* Patients with untreated or uncontrolled hypothyroidism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2018-08-04 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moises Mercado, PhD, Principal Investigator; Aldo Ferreira-Hermosillo, PhD, Principal Investigator — Unafilliated
Locations (1):
- Hospital de Especialidades Centro Médico Nacional Siglo XXI, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon reasonable request to principal investigator

REFERENCES:
- [Background] Barrera-Cruz A, Avila-Jimenez L, Cano-Perez E, Molina-Ayala MA, Parrilla-Ortiz JI, Ramos-Hernandez RI, Sosa-Caballero A, Sosa-Ruiz Mdel R, Gutierrez-Aguilar J. [Practice clinical guideline. Prevention, diagnosis and treatment of overweight and obesity]. Rev Med Inst Mex Seguro Soc. 2013 May-Jun;51(3):344-57. Spanish. PMID 23883468
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] Mason EE, Doherty C, Maher JW, Scott DH, Rodriguez EM, Blommers TJ. Super obesity and gastric reduction procedures. Gastroenterol Clin North Am. 1987 Sep;16(3):495-502. PMID 3436656
- [Background] Nguyen NT, Ho HS, Palmer LS, Wolfe BM. Laparoscopic Roux-en-Y gastric bypass for super/super obesity. Obes Surg. 1999 Aug;9(4):403-6. doi: 10.1381/096089299765553025. PMID 10484302
- [Background] Romero-Martinez M, Shamah-Levy T, Cuevas-Nasu L, Gomez-Humaran IM, Gaona-Pineda EB, Gomez-Acosta LM, Rivera-Dommarco JA, Hernandez-Avila M. [Methodological design of the National Health and Nutrition Survey 2016]. Salud Publica Mex. 2017 May-Jun;59(3):299-305. doi: 10.21149/8593. Spanish. PMID 28902317
- [Background] Barrera-Cruz A, Rodriguez-Gonzalez A, Molina-Ayala MA. [The current state of obesity in Mexico]. Rev Med Inst Mex Seguro Soc. 2013 May-Jun;51(3):292-9. Spanish. PMID 23883458
- [Background] Rizzello M, De Angelis F, Campanile FC, Silecchia G. Effect of gastrointestinal surgical manipulation on metabolic syndrome: a focus on metabolic surgery. Gastroenterol Res Pract. 2012;2012:670418. doi: 10.1155/2012/670418. Epub 2012 Oct 22. PMID 23133447
- [Background] Barquera S, Campos-Nonato I, Hernandez-Barrera L, Pedroza A, Rivera-Dommarco JA. [Prevalence of obesity in Mexican adults 2000-2012]. Salud Publica Mex. 2013;55 Suppl 2:S151-60. Spanish. PMID 24626691
- [Background] Santo MA, Riccioppo D, Pajecki D, Cleva Rd, Kawamoto F, Cecconello I. Preoperative weight loss in super-obese patients: study of the rate of weight loss and its effects on surgical morbidity. Clinics (Sao Paulo). 2014;69(12):828-34. doi: 10.6061/clinics/2014(12)07. PMID 25627995
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S13-S28. doi: 10.2337/dc19-S002. PMID 30559228
- [Background] American Diabetes Association. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S90-S102. doi: 10.2337/dc19-S009. PMID 30559235
- [Background] Apovian CM, Aronne LJ, Bessesen DH, McDonnell ME, Murad MH, Pagotto U, Ryan DH, Still CD; Endocrine Society. Pharmacological management of obesity: an endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2015 Feb;100(2):342-62. doi: 10.1210/jc.2014-3415. Epub 2015 Jan 15. PMID 25590212
- [Background] Yanovski SZ, Yanovski JA. Long-term drug treatment for obesity: a systematic and clinical review. JAMA. 2014 Jan 1;311(1):74-86. doi: 10.1001/jama.2013.281361. PMID 24231879
- [Background] Idris I, Donnelly R. Sodium-glucose co-transporter-2 inhibitors: an emerging new class of oral antidiabetic drug. Diabetes Obes Metab. 2009 Feb;11(2):79-88. doi: 10.1111/j.1463-1326.2008.00982.x. PMID 19125776
- [Background] Shepherd PR, Kahn BB. Glucose transporters and insulin action--implications for insulin resistance and diabetes mellitus. N Engl J Med. 1999 Jul 22;341(4):248-57. doi: 10.1056/NEJM199907223410406. No abstract available. PMID 10413738
- [Background] Wood IS, Trayhurn P. Glucose transporters (GLUT and SGLT): expanded families of sugar transport proteins. Br J Nutr. 2003 Jan;89(1):3-9. doi: 10.1079/BJN2002763. PMID 12568659
- [Background] Oku A, Ueta K, Arakawa K, Ishihara T, Nawano M, Kuronuma Y, Matsumoto M, Saito A, Tsujihara K, Anai M, Asano T, Kanai Y, Endou H. T-1095, an inhibitor of renal Na+-glucose cotransporters, may provide a novel approach to treating diabetes. Diabetes. 1999 Sep;48(9):1794-800. doi: 10.2337/diabetes.48.9.1794. PMID 10480610
- [Background] Ueta K, Ishihara T, Matsumoto Y, Oku A, Nawano M, Fujita T, Saito A, Arakawa K. Long-term treatment with the Na+-glucose cotransporter inhibitor T-1095 causes sustained improvement in hyperglycemia and prevents diabetic neuropathy in Goto-Kakizaki Rats. Life Sci. 2005 Apr 22;76(23):2655-68. doi: 10.1016/j.lfs.2004.09.038. PMID 15792833
- [Background] Meng W, Ellsworth BA, Nirschl AA, McCann PJ, Patel M, Girotra RN, Wu G, Sher PM, Morrison EP, Biller SA, Zahler R, Deshpande PP, Pullockaran A, Hagan DL, Morgan N, Taylor JR, Obermeier MT, Humphreys WG, Khanna A, Discenza L, Robertson JG, Wang A, Han S, Wetterau JR, Janovitz EB, Flint OP, Whaley JM, Washburn WN. Discovery of dapagliflozin: a potent, selective renal sodium-dependent glucose cotransporter 2 (SGLT2) inhibitor for the treatment of type 2 diabetes. J Med Chem. 2008 Mar 13;51(5):1145-9. doi: 10.1021/jm701272q. Epub 2008 Feb 9. PMID 18260618
- [Background] Komoroski B, Vachharajani N, Feng Y, Li L, Kornhauser D, Pfister M. Dapagliflozin, a novel, selective SGLT2 inhibitor, improved glycemic control over 2 weeks in patients with type 2 diabetes mellitus. Clin Pharmacol Ther. 2009 May;85(5):513-9. doi: 10.1038/clpt.2008.250. Epub 2009 Jan 7. PMID 19129749
- [Background] Hussey EK, Dobbins RL, Stoltz RR, Stockman NL, O'Connor-Semmes RL, Kapur A, Murray SC, Layko D, Nunez DJ. Multiple-dose pharmacokinetics and pharmacodynamics of sergliflozin etabonate, a novel inhibitor of glucose reabsorption, in healthy overweight and obese subjects: a randomized double-blind study. J Clin Pharmacol. 2010 Jun;50(6):636-46. doi: 10.1177/0091270009352185. Epub 2010 Mar 3. PMID 20200268
- [Background] Garber AJ, Abrahamson MJ, Barzilay JI, Blonde L, Bloomgarden ZT, Bush MA, Dagogo-Jack S, DeFronzo RA, Einhorn D, Fonseca VA, Garber JR, Garvey WT, Grunberger G, Handelsman Y, Hirsch IB, Jellinger PS, McGill JB, Mechanick JI, Rosenblit PD, Umpierrez GE. CONSENSUS STATEMENT BY THE AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY ON THE COMPREHENSIVE TYPE 2 DIABETES MANAGEMENT ALGORITHM - 2019 EXECUTIVE SUMMARY. Endocr Pract. 2019 Jan;25(1):69-100. doi: 10.4158/CS-2018-0535. No abstract available. PMID 30742570
- [Background] List JF, Woo V, Morales E, Tang W, Fiedorek FT. Sodium-glucose cotransport inhibition with dapagliflozin in type 2 diabetes. Diabetes Care. 2009 Apr;32(4):650-7. doi: 10.2337/dc08-1863. Epub 2008 Dec 29. PMID 19114612
- [Background] Nauck MA, Del Prato S, Duran-Garcia S, Rohwedder K, Langkilde AM, Sugg J, Parikh SJ. Durability of glycaemic efficacy over 2 years with dapagliflozin versus glipizide as add-on therapies in patients whose type 2 diabetes mellitus is inadequately controlled with metformin. Diabetes Obes Metab. 2014 Nov;16(11):1111-20. doi: 10.1111/dom.12327. Epub 2014 Jul 10. PMID 24919526
- [Background] Rosenstock J, Vico M, Wei L, Salsali A, List JF. Effects of dapagliflozin, an SGLT2 inhibitor, on HbA(1c), body weight, and hypoglycemia risk in patients with type 2 diabetes inadequately controlled on pioglitazone monotherapy. Diabetes Care. 2012 Jul;35(7):1473-8. doi: 10.2337/dc11-1693. Epub 2012 Mar 23. PMID 22446170
- [Background] Orme M, Fenici P, Lomon ID, Wygant G, Townsend R, Roudaut M. A systematic review and mixed-treatment comparison of dapagliflozin with existing anti-diabetes treatments for those with type 2 diabetes mellitus inadequately controlled by sulfonylurea monotherapy. Diabetol Metab Syndr. 2014 Jun 11;6:73. doi: 10.1186/1758-5996-6-73. eCollection 2014. PMID 25006351
- [Background] Jabbour SA, Hardy E, Sugg J, Parikh S; Study 10 Group. Dapagliflozin is effective as add-on therapy to sitagliptin with or without metformin: a 24-week, multicenter, randomized, double-blind, placebo-controlled study. Diabetes Care. 2014;37(3):740-50. doi: 10.2337/dc13-0467. Epub 2013 Oct 21. PMID 24144654
- [Background] Fioretto P, Giaccari A, Sesti G. Efficacy and safety of dapagliflozin, a sodium glucose cotransporter 2 (SGLT2) inhibitor, in diabetes mellitus. Cardiovasc Diabetol. 2015 Oct 17;14:142. doi: 10.1186/s12933-015-0297-x. PMID 26474563
- [Background] Dandona P, Mathieu C, Phillip M, Hansen L, Tschope D, Thoren F, Xu J, Langkilde AM; DEPICT-1 Investigators. Efficacy and Safety of Dapagliflozin in Patients With Inadequately Controlled Type 1 Diabetes: The DEPICT-1 52-Week Study. Diabetes Care. 2018 Dec;41(12):2552-2559. doi: 10.2337/dc18-1087. Epub 2018 Oct 23. PMID 30352894
- [Background] Bonner C, Kerr-Conte J, Gmyr V, Queniat G, Moerman E, Thevenet J, Beaucamps C, Delalleau N, Popescu I, Malaisse WJ, Sener A, Deprez B, Abderrahmani A, Staels B, Pattou F. Inhibition of the glucose transporter SGLT2 with dapagliflozin in pancreatic alpha cells triggers glucagon secretion. Nat Med. 2015 May;21(5):512-7. doi: 10.1038/nm.3828. Epub 2015 Apr 20. PMID 25894829
- [Background] Hattersley AT, Thorens B. Type 2 Diabetes, SGLT2 Inhibitors, and Glucose Secretion. N Engl J Med. 2015 Sep 3;373(10):974-6. doi: 10.1056/NEJMcibr1506573. No abstract available. PMID 26332554
- [Background] Saponaro C, Pattou F, Bonner C. SGLT2 inhibition and glucagon secretion in humans. Diabetes Metab. 2018 Nov;44(5):383-385. doi: 10.1016/j.diabet.2018.06.005. Epub 2018 Jun 30. PMID 30017776
- [Background] Liakos A, Karagiannis T, Bekiari E, Boura P, Tsapas A. Update on long-term efficacy and safety of dapagliflozin in patients with type 2 diabetes mellitus. Ther Adv Endocrinol Metab. 2015 Apr;6(2):61-7. doi: 10.1177/2042018814560735. PMID 25941564
- [Background] Baker WL, Smyth LR, Riche DM, Bourret EM, Chamberlin KW, White WB. Effects of sodium-glucose co-transporter 2 inhibitors on blood pressure: a systematic review and meta-analysis. J Am Soc Hypertens. 2014 Apr;8(4):262-75.e9. doi: 10.1016/j.jash.2014.01.007. Epub 2014 Jan 26. PMID 24602971
- [Background] Briasoulis A, Al Dhaybi O, Bakris GL. SGLT2 Inhibitors and Mechanisms of Hypertension. Curr Cardiol Rep. 2018 Jan 19;20(1):1. doi: 10.1007/s11886-018-0943-5. PMID 29349558
- [Background] Jayawardene D, Ward GM, O'Neal DN, Theverkalam G, MacIsaac AI, MacIsaac RJ. New treatments for type 2 diabetes: cardiovascular protection beyond glucose lowering? Heart Lung Circ. 2014 Nov;23(11):997-1008. doi: 10.1016/j.hlc.2014.05.007. Epub 2014 Jun 10. PMID 24996388
- [Background] Hundal RS, Krssak M, Dufour S, Laurent D, Lebon V, Chandramouli V, Inzucchi SE, Schumann WC, Petersen KF, Landau BR, Shulman GI. Mechanism by which metformin reduces glucose production in type 2 diabetes. Diabetes. 2000 Dec;49(12):2063-9. doi: 10.2337/diabetes.49.12.2063. PMID 11118008
- [Background] Pryor R, Cabreiro F. Repurposing metformin: an old drug with new tricks in its binding pockets. Biochem J. 2015 Nov 1;471(3):307-22. doi: 10.1042/BJ20150497. PMID 26475449
- [Background] Goodarzi MO, Bryer-Ash M. Metformin revisited: re-evaluation of its properties and role in the pharmacopoeia of modern antidiabetic agents. Diabetes Obes Metab. 2005 Nov;7(6):654-65. doi: 10.1111/j.1463-1326.2004.00448.x. PMID 16219009
- [Background] Hermann LS, Karlsson JE, Sjostrand A. Prospective comparative study in NIDDM patients of metformin and glibenclamide with special reference to lipid profiles. Eur J Clin Pharmacol. 1991;41(3):263-5. doi: 10.1007/BF00315441. PMID 1748145
- [Background] Stumvoll M, Nurjhan N, Perriello G, Dailey G, Gerich JE. Metabolic effects of metformin in non-insulin-dependent diabetes mellitus. N Engl J Med. 1995 Aug 31;333(9):550-4. doi: 10.1056/NEJM199508313330903. PMID 7623903
- [Background] DeFronzo RA, Goodman AM. Efficacy of metformin in patients with non-insulin-dependent diabetes mellitus. The Multicenter Metformin Study Group. N Engl J Med. 1995 Aug 31;333(9):541-9. doi: 10.1056/NEJM199508313330902. PMID 7623902
- [Background] Mogul HR, Peterson SJ, Weinstein BI, Zhang S, Southren AL. Metformin and carbohydrate-modified diet: a novel obesity treatment protocol: preliminary findings from a case series of nondiabetic women with midlife weight gain and hyperinsulinemia. Heart Dis. 2001 Sep-Oct;3(5):285-92. doi: 10.1097/00132580-200109000-00002. PMID 11975807
- [Background] Devenny JJ, Godonis HE, Harvey SJ, Rooney S, Cullen MJ, Pelleymounter MA. Weight loss induced by chronic dapagliflozin treatment is attenuated by compensatory hyperphagia in diet-induced obese (DIO) rats. Obesity (Silver Spring). 2012 Aug;20(8):1645-52. doi: 10.1038/oby.2012.59. Epub 2012 Mar 8. PMID 22402735
- [Background] Zhang Q, Dou J, Lu J. Combinational therapy with metformin and sodium-glucose cotransporter inhibitors in management of type 2 diabetes: systematic review and meta-analyses. Diabetes Res Clin Pract. 2014 Sep;105(3):313-21. doi: 10.1016/j.diabres.2014.06.006. Epub 2014 Jun 22. PMID 25015317
- [Background] Nowak A, Czkwianianc E. A contemporary approach to body mass regulation mechanisms. Prz Gastroenterol. 2016;11(2):73-7. doi: 10.5114/pg.2016.60043. Epub 2016 May 19. PMID 27350833
- [Background] Bolinder J, Ljunggren O, Kullberg J, Johansson L, Wilding J, Langkilde AM, Sugg J, Parikh S. Effects of dapagliflozin on body weight, total fat mass, and regional adipose tissue distribution in patients with type 2 diabetes mellitus with inadequate glycemic control on metformin. J Clin Endocrinol Metab. 2012 Mar;97(3):1020-31. doi: 10.1210/jc.2011-2260. Epub 2012 Jan 11. PMID 22238392
- [Background] Gregor MF, Hotamisligil GS. Inflammatory mechanisms in obesity. Annu Rev Immunol. 2011;29:415-45. doi: 10.1146/annurev-immunol-031210-101322. PMID 21219177
- [Background] Fernandez-Sanchez A, Madrigal-Santillan E, Bautista M, Esquivel-Soto J, Morales-Gonzalez A, Esquivel-Chirino C, Durante-Montiel I, Sanchez-Rivera G, Valadez-Vega C, Morales-Gonzalez JA. Inflammation, oxidative stress, and obesity. Int J Mol Sci. 2011;12(5):3117-32. doi: 10.3390/ijms12053117. Epub 2011 May 13. PMID 21686173
- [Background] Hajer GR, van Haeften TW, Visseren FL. Adipose tissue dysfunction in obesity, diabetes, and vascular diseases. Eur Heart J. 2008 Dec;29(24):2959-71. doi: 10.1093/eurheartj/ehn387. Epub 2008 Sep 5. PMID 18775919
- [Background] Kalupahana NS, Moustaid-Moussa N, Claycombe KJ. Immunity as a link between obesity and insulin resistance. Mol Aspects Med. 2012 Feb;33(1):26-34. doi: 10.1016/j.mam.2011.10.011. Epub 2011 Oct 21. PMID 22040698
- [Background] Wang Z, Nakayama T. Inflammation, a link between obesity and cardiovascular disease. Mediators Inflamm. 2010;2010:535918. doi: 10.1155/2010/535918. Epub 2010 Aug 5. PMID 20847813
- [Background] Wolf G. Serum retinol-binding protein: a link between obesity, insulin resistance, and type 2 diabetes. Nutr Rev. 2007 May;65(5):251-6. doi: 10.1111/j.1753-4887.2007.tb00302.x. PMID 17566551
- [Background] Bluher M, Fasshauer M, Tonjes A, Kratzsch J, Schon MR, Paschke R. Association of interleukin-6, C-reactive protein, interleukin-10 and adiponectin plasma concentrations with measures of obesity, insulin sensitivity and glucose metabolism. Exp Clin Endocrinol Diabetes. 2005 Oct;113(9):534-7. doi: 10.1055/s-2005-872851. PMID 16235156
- [Background] Patel PS, Buras ED, Balasubramanyam A. The role of the immune system in obesity and insulin resistance. J Obes. 2013;2013:616193. doi: 10.1155/2013/616193. Epub 2013 Mar 21. PMID 23577240
- [Background] Queipo-Ortuno MI, Escote X, Ceperuelo-Mallafre V, Garrido-Sanchez L, Miranda M, Clemente-Postigo M, Perez-Perez R, Peral B, Cardona F, Fernandez-Real JM, Tinahones FJ, Vendrell J. FABP4 dynamics in obesity: discrepancies in adipose tissue and liver expression regarding circulating plasma levels. PLoS One. 2012;7(11):e48605. doi: 10.1371/journal.pone.0048605. Epub 2012 Nov 5. PMID 23139800
- [Background] Goktas Z, Moustaid-Moussa N, Shen CL, Boylan M, Mo H, Wang S. Effects of bariatric surgery on adipokine-induced inflammation and insulin resistance. Front Endocrinol (Lausanne). 2013 Jun 10;4:69. doi: 10.3389/fendo.2013.00069. eCollection 2013. PMID 23772224
- [Background] Weisberg SP, McCann D, Desai M, Rosenbaum M, Leibel RL, Ferrante AW Jr. Obesity is associated with macrophage accumulation in adipose tissue. J Clin Invest. 2003 Dec;112(12):1796-808. doi: 10.1172/JCI19246. PMID 14679176
- [Background] Garcia de la Torre N, Rubio MA, Bordiu E, Cabrerizo L, Aparicio E, Hernandez C, Sanchez-Pernaute A, Diez-Valladares L, Torres AJ, Puente M, Charro AL. Effects of weight loss after bariatric surgery for morbid obesity on vascular endothelial growth factor-A, adipocytokines, and insulin. J Clin Endocrinol Metab. 2008 Nov;93(11):4276-81. doi: 10.1210/jc.2007-1370. Epub 2008 Aug 19. PMID 18713823
- [Background] Leick L, Lindegaard B, Stensvold D, Plomgaard P, Saltin B, Pilegaard H. Adipose tissue interleukin-18 mRNA and plasma interleukin-18: effect of obesity and exercise. Obesity (Silver Spring). 2007 Feb;15(2):356-63. doi: 10.1038/oby.2007.528. PMID 17299108
- [Background] Panee J. Monocyte Chemoattractant Protein 1 (MCP-1) in obesity and diabetes. Cytokine. 2012 Oct;60(1):1-12. doi: 10.1016/j.cyto.2012.06.018. Epub 2012 Jul 4. PMID 22766373
- [Background] Okamoto A, Yokokawa H, Sanada H, Naito T. Changes in Levels of Biomarkers Associated with Adipocyte Function and Insulin and Glucagon Kinetics During Treatment with Dapagliflozin Among Obese Type 2 Diabetes Mellitus Patients. Drugs R D. 2016 Sep;16(3):255-261. doi: 10.1007/s40268-016-0137-9. PMID 27333994
- [Background] Steppan CM, Bailey ST, Bhat S, Brown EJ, Banerjee RR, Wright CM, Patel HR, Ahima RS, Lazar MA. The hormone resistin links obesity to diabetes. Nature. 2001 Jan 18;409(6818):307-12. doi: 10.1038/35053000. PMID 11201732
- [Background] Tilg H, Moschen AR. Role of adiponectin and PBEF/visfatin as regulators of inflammation: involvement in obesity-associated diseases. Clin Sci (Lond). 2008 Feb;114(4):275-88. doi: 10.1042/CS20070196. PMID 18194136
- [Background] Vidal-Puig A, O'Rahilly S. Resistin: a new link between obesity and insulin resistance? Clin Endocrinol (Oxf). 2001 Oct;55(4):437-8. doi: 10.1046/j.1365-2265.2001.01377.x. No abstract available. PMID 11678824
- [Background] Fernandez-Real JM, Vayreda M, Richart C, Gutierrez C, Broch M, Vendrell J, Ricart W. Circulating interleukin 6 levels, blood pressure, and insulin sensitivity in apparently healthy men and women. J Clin Endocrinol Metab. 2001 Mar;86(3):1154-9. doi: 10.1210/jcem.86.3.7305. PMID 11238501
- [Background] Senn JJ, Klover PJ, Nowak IA, Mooney RA. Interleukin-6 induces cellular insulin resistance in hepatocytes. Diabetes. 2002 Dec;51(12):3391-9. doi: 10.2337/diabetes.51.12.3391. PMID 12453891
- [Background] Steinberg GR. Inflammation in obesity is the common link between defects in fatty acid metabolism and insulin resistance. Cell Cycle. 2007 Apr 15;6(8):888-94. doi: 10.4161/cc.6.8.4135. Epub 2007 Apr 11. PMID 17438370
- [Background] Moore KW, de Waal Malefyt R, Coffman RL, O'Garra A. Interleukin-10 and the interleukin-10 receptor. Annu Rev Immunol. 2001;19:683-765. doi: 10.1146/annurev.immunol.19.1.683. PMID 11244051
- [Background] Hotamisligil GS, Shargill NS, Spiegelman BM. Adipose expression of tumor necrosis factor-alpha: direct role in obesity-linked insulin resistance. Science. 1993 Jan 1;259(5091):87-91. doi: 10.1126/science.7678183.
- [Background] Kanety H, Feinstein R, Papa MZ, Hemi R, Karasik A. Tumor necrosis factor alpha-induced phosphorylation of insulin receptor substrate-1 (IRS-1). Possible mechanism for suppression of insulin-stimulated tyrosine phosphorylation of IRS-1. J Biol Chem. 1995 Oct 6;270(40):23780-4. doi: 10.1074/jbc.270.40.23780. PMID 7559552
- [Background] Warne JP. Tumour necrosis factor alpha: a key regulator of adipose tissue mass. J Endocrinol. 2003 Jun;177(3):351-5. doi: 10.1677/joe.0.1770351. PMID 12773114
- [Background] Vasilakou D, Karagiannis T, Athanasiadou E, Mainou M, Liakos A, Bekiari E, Sarigianni M, Matthews DR, Tsapas A. Sodium-glucose cotransporter 2 inhibitors for type 2 diabetes: a systematic review and meta-analysis. Ann Intern Med. 2013 Aug 20;159(4):262-74. doi: 10.7326/0003-4819-159-4-201308200-00007. PMID 24026259
- [Background] Kelly MS, Lewis J, Huntsberry AM, Dea L, Portillo I. Efficacy and renal outcomes of SGLT2 inhibitors in patients with type 2 diabetes and chronic kidney disease. Postgrad Med. 2019 Jan;131(1):31-42. doi: 10.1080/00325481.2019.1549459. Epub 2018 Nov 30. PMID 30449220
- [Background] Rosenstock J, Ferrannini E. Euglycemic Diabetic Ketoacidosis: A Predictable, Detectable, and Preventable Safety Concern With SGLT2 Inhibitors. Diabetes Care. 2015 Sep;38(9):1638-42. doi: 10.2337/dc15-1380. No abstract available. PMID 26294774
- [Background] Peters AL, Buschur EO, Buse JB, Cohan P, Diner JC, Hirsch IB. Euglycemic Diabetic Ketoacidosis: A Potential Complication of Treatment With Sodium-Glucose Cotransporter 2 Inhibition. Diabetes Care. 2015 Sep;38(9):1687-93. doi: 10.2337/dc15-0843. Epub 2015 Jun 15. PMID 26078479
- [Background] Handelsman Y, Henry RR, Bloomgarden ZT, Dagogo-Jack S, DeFronzo RA, Einhorn D, Ferrannini E, Fonseca VA, Garber AJ, Grunberger G, LeRoith D, Umpierrez GE, Weir MR. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY POSITION STATEMENT ON THE ASSOCIATION OF SGLT-2 INHIBITORS AND DIABETIC KETOACIDOSIS. Endocr Pract. 2016 Jun;22(6):753-62. doi: 10.4158/EP161292.PS. Epub 2016 Jun 1. PMID 27082665
- [Background] Monami M, Nreu B, Zannoni S, Lualdi C, Mannucci E. Effects of SGLT-2 inhibitors on diabetic ketoacidosis: A meta-analysis of randomised controlled trials. Diabetes Res Clin Pract. 2017 Aug;130:53-60. doi: 10.1016/j.diabres.2017.04.017. Epub 2017 May 18. PMID 28570924
- [Background] Erondu N, Desai M, Ways K, Meininger G. Diabetic Ketoacidosis and Related Events in the Canagliflozin Type 2 Diabetes Clinical Program. Diabetes Care. 2015 Sep;38(9):1680-6. doi: 10.2337/dc15-1251. Epub 2015 Jul 22. PMID 26203064
- [Background] Scheen AJ. An update on the safety of SGLT2 inhibitors. Expert Opin Drug Saf. 2019 Apr;18(4):295-311. doi: 10.1080/14740338.2019.1602116. Epub 2019 Apr 16. PMID 30933547
- [Background] Ferrannini E, Muscelli E, Frascerra S, Baldi S, Mari A, Heise T, Broedl UC, Woerle HJ. Metabolic response to sodium-glucose cotransporter 2 inhibition in type 2 diabetic patients. J Clin Invest. 2014 Feb;124(2):499-508. doi: 10.1172/JCI72227. Epub 2014 Jan 27. PMID 24463454
- [Background] Luzi L, Barrett EJ, Groop LC, Ferrannini E, DeFronzo RA. Metabolic effects of low-dose insulin therapy on glucose metabolism in diabetic ketoacidosis. Diabetes. 1988 Nov;37(11):1470-7. doi: 10.2337/diab.37.11.1470. PMID 3141236
- [Background] Nogues Solan X, Sorli Redo ML, Villar Garcia J. [Tools to measure treatment adherence]. An Med Interna. 2007 Mar;24(3):138-41. doi: 10.4321/s0212-71992007000300009. Spanish. PMID 17590137
- [Background] Furtado RHM, Bonaca MP, Raz I, Zelniker TA, Mosenzon O, Cahn A, Kuder J, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Nicolau JC, Gause-Nilsson IAM, Fredriksson M, Langkilde AM, Sabatine MS, Wiviott SD. Dapagliflozin and Cardiovascular Outcomes in Patients With Type 2 Diabetes Mellitus and Previous Myocardial Infarction. Circulation. 2019 May 28;139(22):2516-2527. doi: 10.1161/CIRCULATIONAHA.119.039996. Epub 2019 Mar 18. PMID 30882239
- [Background] Wilding J, Bailey C, Rigney U, Blak B, Beekman W, Emmas C. Glycated Hemoglobin, Body Weight and Blood Pressure in Type 2 Diabetes Patients Initiating Dapagliflozin Treatment in Primary Care: A Retrospective Study. Diabetes Ther. 2016 Dec;7(4):695-711. doi: 10.1007/s13300-016-0193-8. Epub 2016 Sep 1. PMID 27585582
- [Background] Schork A, Saynisch J, Vosseler A, Jaghutriz BA, Heyne N, Peter A, Haring HU, Stefan N, Fritsche A, Artunc F. Effect of SGLT2 inhibitors on body composition, fluid status and renin-angiotensin-aldosterone system in type 2 diabetes: a prospective study using bioimpedance spectroscopy. Cardiovasc Diabetol. 2019 Apr 5;18(1):46. doi: 10.1186/s12933-019-0852-y. PMID 30953516
- [Background] Calapkulu M, Cander S, Gul OO, Ersoy C. Anthropometric outcomes in type 2 diabetic patients with new dapagliflozin treatment; actual clinical experience data of six months retrospective glycemic control from single center. Diabetes Metab Syndr. 2019 Jan-Feb;13(1):284-288. doi: 10.1016/j.dsx.2018.09.005. Epub 2018 Sep 8. PMID 30641713
- [Background] Faerch K, Amadid H, Nielsen LB, Ried-Larsen M, Karstoft K, Persson F, Jorgensen ME. Protocol for a randomised controlled trial of the effect of dapagliflozin, metformin and exercise on glycaemic variability, body composition and cardiovascular risk in prediabetes (the PRE-D Trial). BMJ Open. 2017 Jun 6;7(5):e013802. doi: 10.1136/bmjopen-2016-013802. PMID 28592573
- [Derived] Ferreira-Hermosillo A, Molina-Ayala MA, Molina-Guerrero D, Garrido-Mendoza AP, Ramirez-Renteria C, Mendoza-Zubieta V, Espinosa E, Mercado M. Efficacy of the treatment with dapagliflozin and metformin compared to metformin monotherapy for weight loss in patients with class III obesity: a randomized controlled trial. Trials. 2020 Feb 14;21(1):186. doi: 10.1186/s13063-020-4121-x. PMID 32059692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with grade III obesity undergoing a bariatric surgery protocol were recluded at Hospital de Especialidades Centro Medico Nacional Siglo XXI, IMSS between 2018 and 2024. The first participant was enrolled on August 4th 2018 and the last participant was enrolled in July 31st 2023.
Pre-assignment Details: Of 160 enrolled participants, 109 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | Metformin/Dapagliflozin | Metformin
Started | 54 | 55
Completed | 43 | 37
Not Completed | 11 | 18
Not completed — Lost to Follow-up | 11 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin/Dapagliflozin | Metformin | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Customized [Mean (Standard Deviation); unit: years] — Time elapsed from birth to the present (18-60 years)
  years
    Years | 46 (8) | 42 (9) | 44 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 18 | 17 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 55 | 109
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Mexico
  participants
    Mexico | 54 | 55 | 109

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Change in weight using (dapaglifozin/metformin) vs. metformin at one, three, six, nine and twelve months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Metformin/Dapagliflozin: Metformin 1,700 mg/day and Dapagliflozin 10 mg/day for a year.
  Dapagliflozin/Metformin: Two tablets of Metformin 850 mg every 12 hours will be provided in combination with Dapagliflozin 10 mg per day. Each participant will receive diet and exercise intervention according to their BMI and current physical condition.
- Metformin: Metformin 1,700 mg/day
  Metformin: Two tablets of Metformin 850 mg every 12 hours will be provided. Each participant will receive diet and exercise intervention according to their BMI and current physical condition.
Arm/Group | Metformin/Dapagliflozin | Metformin
Number analyzed (Participants) | 54 | 55
kg
  Initial weight | 121.5 (21.1) | 125.9 (23.9)
  Weight (1 month) | 118 (20.8) | 123.7 (21.8)
  Weight (3 months) | 116.3 (20.11) | 120 (20.58)
  Weight (6 months) | 114.4 (17.8) | 119.9 (22.4)
  Weight (9 months) | 115.4 (17.9) | 118.4 (21.4)
  Final weight (12 months) | 116 (19) | 115 (20.18)
Statistical Analysis 1: Comparison: Metformin/Dapagliflozin vs Metformin; Test type: Superiority; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Change in Blood Pressure
Description: Change in blood pressure using (dapaglifozin/metformin) vs. metformin at three, six, nine and twelve months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Metformin/Dapagliflozin | Metformin
Number analyzed (Participants) | 54 | 55
mmHg
  Initial Systolic blood pressure | 115 (14) | 120 (13)
  Initial Diastolic blood pressure | 80 (10) | 81 (8)
  Systolic blood pressure (3 months) | 113 (14) | 199 (11)
  Diastolic blood pressure (3 months) | 77 (9) | 78 (13)
  Systolic blood pressure (6 months) | 113 (11) | 118 (15)
  Diastolic blood pressure (6 months) | 77 (8) | 78 (9)
  Systolic blood pressure (9 months) | 114 (14) | 116 (13)
  Diastolic blood pressure (9 months) | 77 (11) | 74 (8)
  Final Systolic blood pressure (12 months) | 122 (14) | 120 (20)
  Final Diastolic blood pressure (12 months) | 79 (8) | 76 (8)
Statistical Analysis 1: Comparison: Metformin/Dapagliflozin vs Metformin; Test type: Other; p < 0.05, Mixed Models Analysis

3. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference in (dapaglifozin/metformin) vs. metformin at one, three, six, nine and twelve months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Metformin/Dapagliflozin | Metformin
Number analyzed (Participants) | 54 | 55
cm
  Initial waist circumference | 130 (13) | 131 (14)
  Waist circumference (1 month) | 123 (22) | 129 (11)
  Waist circumference (3 months) | 124 (14) | 126 (13)
  Waist circumference (6 months) | 124 (12) | 124 (13)
  Waist circumference (9 months) | 124 (11) | 124 (14)
  Final waist circumference ( 12 months) | 125 (11) | 123 (11)
Statistical Analysis 1: Comparison: Metformin/Dapagliflozin vs Metformin; Test type: Other; p < 0.05, Mixed Models Analysis

4. Secondary Outcome: Change in Lipid Levels
Description: Change in lipid levels using (dapaglifozin/metformin) vs. metformin in three, six, nine and twelve months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Metformin/Dapagliflozin | Metformin
Number analyzed (Participants) | 54 | 55
mg/dl
  Initial c-HDL | 41 (10) | 39 (8)
  Initial c-LDL | 91 (27) | 93 (29)
  Initial CT | 167 (29) | 162 (33)
  Initial TAG | 154 (122) | 138 (107)
  c-HDL (3 months) | 42 (9) | 41 (9)
  c-LDL (3 months) | 89 (27) | 41 (9)
  CT (3 months) | 161 (39) | 164 (32)
  TAG (3 months) | 158 (117) | 154 (111)
  c-HDL (6 months) | 42 (10) | 42 (9)
  c-LDL (6 months) | 93 (27) | 42 (9)
  CT (6 months) | 167 (30) | 173 (31)
  TAG (6 months) | 146 (116) | 142 (131)
  c-HDL (9 months) | 49 (19) | 43 (9)
  c-LDL (9 months) | 98 (36) | 43 (9)
  CT (9 months) | 174 (41) | 168 (40)
  TAG (9 months) | 145 (124) | 136 (114)
  Final c-HDL (12 months) | 42 (10) | 43 (9)
  Final c-LDL (12 months) | 96 (29) | 94 (22)
  Final CT (12 months) | 173 (42) | 168 (24)
  Final TAG (12 months) | 145 (122) | 154 (122)
Statistical Analysis 1: Comparison: Metformin/Dapagliflozin vs Metformin; Test type: Other; p < 0.05, Mixed Models Analysis

5. Other Pre Specified Outcome: Change in Cytokines Level
Description: Change in cytokines using (dapaglifozin/metformin) vs. metformin.
Time Frame: 12 months
Measure: Mean (Inter-Quartile Range); unit: pg/ml
Arm/Group | Metformin/Dapagliflozin | Metformin
Number analyzed (Participants) | 54 | 55
pg/ml
  Initial IL-10 | 6.34 [2.44 to 17.67] | 3.09 [1.66 to 13.29]
  Initial IL-6 | 13.89 [6.81 to 46.6] | 9.16 [4.36 to 20.26]
  Initial TNF-alfa | 16.85 [11.68 to 20.94] | 11.34 [8.61 to 14.44]
  Initial Resistin | 2468.2 [1912.7 to 3245.6] | 2503.75 [1707.6 to 3691.3]
  Final IL-10 (12 months) | 8.46 [2.9 to 28.4] | 4.06 [1.66 to 8.35]
  Final IL-6 (12 months) | 15.69 [6.71 to 56.8] | 6.43 [4.38 to 23.65]
  Final TNF-alfa (12 months) | 16.59 [11.55 to 23.11] | 10.02 [8.35 to 13.46]
  Final resistin (12 months) | 2468.2 [1912.7 to 3245.6] | 2344.98 [1925.6 to 3263.47]

6. Other Pre Specified Outcome: Change in Adiponectin
Description: Change in adiponectin using (dapaglifozin/metformin) vs. metformin.
Time Frame: 12 months
Measure: Mean (Inter-Quartile Range); unit: ng/ml
Arm/Group | Metformin/Dapagliflozin | Metformin
Number analyzed (Participants) | 54 | 55
ng/ml
  Initial Adiponectin | 68604.3 [43943.1 to 102091] | 49880.4 [35824.5 to 73390.2]
  Final adiponectin (12 months) | 77119.2 [59033.8 to 96640.6] | 63587.4 [39261.4 to 81996.9]

7. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change in body mass index (dapaglifozin/metformin) vs. metformin at one, three, six, nine and twelve months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Metformin/Dapagliflozin | Metformin
Number analyzed (Participants) | 54 | 55
kg/m2
  Initial BMI | 45.2 (42.3) | 45.6 (43.2)
  BMI (1 month) | 44.1 (41.2) | 45.4 (42.5)
  BMI (3 months) | 43.5 (40.3) | 44.4 (41.5)
  BMI (6 months) | 43.1 (40.6) | 43.7 (40.6)
  BMI (9 months) | 43.3 (41.6) | 43.3 (40.5)
  Final BMI (12 months) | 44.4 (41.4) | 42.9 (39.5)

ADVERSE EVENTS:
Time Frame: 12 months.
Arm/Group | Metformin/Dapagliflozin | Metformin
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/55
Other Adverse Events (participants affected / at risk) | 15/54 | 8/55
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin/Dapagliflozin (N=54) | Metformin (N=55)
Genital Tract Infections (Infections and infestations) | 15 (15) | 8 (8)

LIMITATIONS AND CAVEATS:
Delay in the study completion due COVID-19 pandemic. We were not able to measure glucagon and ghrelin concentrations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT03968224/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT03968224/ICF_001.pdf